CLINICAL TRIAL: NCT06201013
Title: Efficacy and Safety of Vitamin D in the Treatment of Wet Overactive Bladder in Children: a Clinical Randomized Controlled Test
Brief Title: Efficacy and Safety of Vitamin D in the Treatment of OAB-wet in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xing Liu (Other)
Responsible Party: Sponsor-Investigator, Xing Liu, Professor, Doctor, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023922
Record Dates: First submitted 2023-09-26; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-09

CONDITIONS: Urinary Bladder, Overactive; Overactive Bladder; Urinary Incontinence, Urge
Keywords: Urinary Bladder, Overactive; Urinary Incontinence, Urge; Vitamin D
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge | interventions — Solifenacin Succinate; Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Urotherapy (Placebo Comparator): Participants were asked to undergo a 30-minute course every 6 weeks at follow-up, including (1) education to dispel doubts about the disease and understand the benefits of curing dysfunction to facilitate better treatment outcomes for children, (2) regular urination to establish good urination habits, (3) dietary guidance to avoid constipation, and (4) how to accurately record symptoms of OAB
  Interventions: Behavioral: urotherapy
- Standard Urotherapy Combined with Solifenacin Drug Treatment (Active Comparator): Standard Urotherapy plus Solinasine succinate 5mg once daily with a maximum dose of 10mg/day
  Interventions: Behavioral: urotherapy; Drug: Solifenacin Succinate
- Standard Urotherapy Combined with Vitamin D supplementation (Experimental): Standard Urotherapy plus high dose vitamin D supplement 2400iu/d
  Interventions: Behavioral: urotherapy; Drug: Vitamin D3

INTERVENTIONS:
Behavioral: urotherapy — Participants were asked to undergo a 30-min session every 6 weeks at follow-up, including (1) education about the disease to dispel doubts about it and to understand the benefits of curing the dysfunction in order for the child to have a better therapeutic outcome, (2) urination at regular intervals and the establishment of good urination habits, (3) dietary instructions to avoid constipation, (4) accurate recording of symptoms of OAB, and (5) communication with the research team every 2 weeks.
Drug: Solifenacin Succinate — In addition to urotherapy, take Solifenacin succinate 5mg once daily, maximum dose 10 mg/day
  Other Names: andard Urotherapy Combined with Solifenacin Drug Treatment
  Arms: Standard Urotherapy Combined with Solifenacin Drug Treatment
Drug: Vitamin D3 — In addition to urologic therapy, vitamin D drops containing 400 IU of vitamin D3 per capsule, 1,200 iu per oral dose, twice daily, for a total of 2,400 iu/d; serum vitamin D levels need to be rechecked at every 6-week follow-up visit
  Other Names: Standard Urotherapy Combined with Vitamin D supplementation
  Arms: Standard Urotherapy Combined with Vitamin D supplementation

SUMMARY:
The purpose of this clinical trial is to investigate whether standard behavioral therapy combined with high-dose vitamin D (2400iu daily) is superior to standard behavioral therapy alone and standard behavioral therapy combined with solifenacin medication in improving frequency of incontinence and lower urinary tract symptom scores in children with wet OAB. Dedicated to understanding the current best treatment for wet OAB and to informing future clinical decisions and improving patient prognosis. The main questions it seeks to answer are

* Question 1 To attempt to elucidate the relationship between vitamin D levels and their lower urinary tract symptoms.
* Question 2 To examine the etiologic role of vitamin D in wet OAB in children.
* Question 3 Compare the effectiveness and safety of interventions to elucidate the etiologic mechanisms and optimal intervention strategies for wet OAB in children.

The researchers will compare (1) standard behavioral therapy with solifenacin (2) standard behavioral therapy with high-dose vitamin D (3) standard behavioral therapy alone to observe the clinical efficacy and safety of the three interventions for children with wet OAB.

DETAILED DESCRIPTION:
[Study Objective]. Primary objective: to investigate whether standard behavioral therapy combined with high-dose vitamin D (2400iu per day) is superior to standard behavioral therapy alone and standard behavioral therapy combined with solifenacin medication in improving frequency of urinary incontinence and lower urinary tract symptom scores in children with wet OAB.

Secondary objectives:

1. To investigate whether this standard behavioral therapy combined with oral solifenacin and vitamin D supplementation regimen is superior to the remaining two groups in the following secondary efficacy outcomes.

   * Number of urinations per day
   * number of nocturia
   * Quality of life
   * Serum vitamin D levels
   * Overall patient satisfaction with treatment
2. To examine whether any effect of vitamin D supplementation on the above outcomes is modified by baseline vitamin D levels, and baseline lower urinary tract symptom severity (secondary outcome, efficacy).
3. Explore whether the treatment regimen of standard behavioral therapy combined with oral solifenacin and vitamin D is safe and well tolerated (secondary outcome, safety).

[Study Steps].

1. Design of Randomization Methods: After completion of a comprehensive baseline assessment, eligible participants are randomized 1:1:1 into three distinct intervention groups. Statisticians independent of this clinical monitoring will generate a randomization table from the PROC PLAN process of the SAS program based on predetermined seed and block numbers. The generated randomization codes will be recorded sequentially in sealed envelopes entrusted to the custody of the residents not involved in the trial.
2. Procedure for inclusion of study subjects: participants will be selected among patients with confirmed wet OAB and serum vitamin D levels below 35 ng/ml in the urology department of our hospital. We will exclude patients with other organic diseases and poor compliance. The guardians of the children will obtain informed consent and sign a paper consent form before starting the intervention.

4.Clinical data collection: information on the demographic characteristics of the child at the initial visit, medical history, family history, history of maternal vitamin D supplementation during pregnancy, history of vitamin D supplementation in the child, laboratory findings (serum vitamin D, routine urinalysis), abdominal imaging findings, and a diary of voiding will be kept by the participant for 7 days to establish a baseline.

ELIGIBILITY:
Inclusion Criteria:

* Children older than or equal to 5 years of age with a diagnosis of wet OAB (the diagnosis followed the latest guidelines of ICCS) attending the outpatient clinic of the Department of Urology of the Affiliated Children's Hospital of Chongqing Medical University,
* children with serum vitamin D levels below 35 ng/ml as indicated by the tests conducted by the hospital
* children whose guardians have given their informed consent, are able to ensure compliance and have signed a paper-based informed consent form.

Exclusion Criteria:

* Those with urinary malformations or serious diseases (e.g., hypospadias, cryptorchidism, posterior urethral valvulae, vesicoureteral reflux, neurogenic bladder, urinary tumors, urinary stones, bladder and urethral injuries, etc.)
* Those with neurological disorders (e.g., epilepsy, spinal cord injuries, spinal dysplasia, spinal embolism syndrome, multiple sclerosis, and autism spectrum disorders, etc.)
* People with serious heart disease, abnormal liver and kidney function, lung disease, bone deformity, serious digestive tract disease, genetic metabolic disease
* People with history of gastrointestinal surgery and urological surgery
* People with dry stools and long-term constipation
* People who are taking anticonvulsant and antiepileptic drugs, hormones, and anti-tuberculosis drugs
* People with history of hypercalcemia, hyperphosphatemia with renal rickets
* People who have had unexplained hematuria and hematuria with renal rickets within the last year
* People who have been suffering from severe heart disease or chronic diabetes.
* participation in other clinical studies at the time of consultation or during the follow-up period of other clinical studies
* unwillingness to participate in this study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-03 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
urinary incontinence frequency | week 1, week6，week 12
  The number of daily occurrences of incontinence recorded through a bladder diary
Lower urinary tract symptom score | week 1, week6，week 12
  Lower urinary tract symptom scale score

SECONDARY OUTCOMES:
Frequency of urination per day | week 1, week6，week 12
  Record the daily frequency of urination using a voiding diary
Qol score | week 1, week6，week 12
  Quality of life was investigated by questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China